CLINICAL TRIAL: NCT00005257
Title: Diet and Plasma Cholesterol - Secular Trend Analysis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1139; R01HL043919 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypercholesterolemia

SUMMARY:
To define the role of dietary variables on changes in plasma cholesterol levels over time in the Framingham cohort and the Framingham Offspring cohort.

DETAILED DESCRIPTION:
BACKGROUND:

Mortality from coronary heart disease has declined over 40 percent since the late 1960s. Possible explanations for the decline include the observed trends in risk factors such as changes in rates of hypertension, dyslipidemia, and glucose intolerance; lifestyle changes such as improvements in diet and decreases in the levels of cigarette smoking; and better detection and treatment of heart disease. The specific effects of risk factor, lifestyle, or detection and treatment changes on the declining population rates of coronary heart disease morbidity and mortality were unknown in 1990. Secular trend analyses were needed to elucidate the relative contribution of these factors, particularly dietary variables, on population rates of coronary heart disease.

DESIGN NARRATIVE:

Multiple regression was used to assess the effect of dietary variables on changes in serum cholesterol between 1957-1960 and 1966-1969 in a sample of 200 men for whom repeated measurements existed in the Framingham cohort. Analysis of covariance was used to assess influence of dietary intake on differences in serum cholesterol levels between independent samples of men studied in 1957-1960 and 1966-1969 in the Framingham cohort, and independent samples of women studied between 1957-1960 and 1984-1988 in the Framingham cohort and Offspring cohort, and independent samples of men studied between 1966-1969 and 1984-1988 in the Framingham cohort and Offspring cohorts respectively.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-05; Study Completion 1992-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Posner — Boston University

REFERENCES:
- [Background] Campos H, Willett WC, Peterson RM, Siles X, Bailey SM, Wilson PW, Posner BM, Ordovas JM, Schaefer EJ. Nutrient intake comparisons between Framingham and rural and Urban Puriscal, Costa Rica. Associations with lipoproteins, apolipoproteins, and low density lipoprotein particle size. Arterioscler Thromb. 1991 Jul-Aug;11(4):1089-99. doi: 10.1161/01.atv.11.4.1089. PMID 2065030
- [Background] Posner BM, Franz MM, Quatromoni PA, Gagnon DR, Sytkowski PA, D'Agostino RB, Cupples LA. Secular trends in diet and risk factors for cardiovascular disease: the Framingham Study. J Am Diet Assoc. 1995 Feb;95(2):171-9. doi: 10.1016/S0002-8223(95)00043-7. PMID 7852683